CLINICAL TRIAL: NCT02696681
Title: Addressing Psychosocial Comorbidities in HIV Treatment and Prevention: Phase 2
Brief Title: Addressing Psychosocial Comorbidities in HIV Treatment and Prevention
Acronym: APPROACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steven Safren, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20150383; 1K24MH094214-01 (NIH); 9K24DA040489-07 (NIH)
Record Dates: First submitted 2016-02-18; First posted 2016-03-02 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Human Immunodeficiency Virus; Depression; Mental Health
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression; Psychological Well-Being | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive Behavioral Therapy (Experimental): Integrating CBT for any substance use or mental health problems with CBT for adherence/self-care
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Integrating CBT for mental health and substance issues concern with CBT for health behavior change

SUMMARY:
Project AProaCH is an open pilot trial of a cognitive behavioral therapy (CBT) for individuals with HIV with various psychological comorbidities, which the investigators call "syndemics". Syndemics are co-occurring psychosocial problems that interact with each other and with health behavior such as HIV sexual transmission risk behavior and adherence to self care.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ individuals
* Uncontrolled virus (plasma HIV RNA concentrations that reach detectable limits) or being diagnosed with a sexually transmitted infection (STI) (gonorrhea, chlamydia, syphilis, trichomoniasis (female only)) currently or within the past 3 months.

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Active untreated, unstable, major mental illness (i.e., untreated psychosis or mania) that would interfere with study participation
* Opinion of the PI that the participant would be at risk for harm to himself or others as a result of study participation,
* Under the age of 18 or over the age of 65,
* Current CBT for a psychiatric disorder, or a course of CBT in the past year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Responder status as defined by the number of participants who change from a detectable to suppressed (undetectable) HIV viral load | 4 months assessment
  Attaining viral suppression
Responder status as defined by the number of participants who change from a detectable to suppressed (undetectable) HIV viral load | 8 month assessment
  Attaining viral suppression

SECONDARY OUTCOMES:
Adherence to antiretroviral therapy via real time monitoring | Changes over time from baseline to 8 month follow-up
  Adherence to ART will be measured using a real time monitoring devices that tracks when a pill box is opened and closed.

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Safren, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Derived] Safren SA, Harkness A, Lee JS, Rogers BG, Mendez NA, Magidson JF, Blashill AJ, Bainter S, Rodriguez A, Ironson G. Addressing Syndemics and Self-care in Individuals with Uncontrolled HIV: An Open Trial of a Transdiagnostic Treatment. AIDS Behav. 2020 Nov;24(11):3264-3278. doi: 10.1007/s10461-020-02900-7. PMID 32410049